CLINICAL TRIAL: NCT02416232
Title: An Open Label Non Randomized Access Study of Trametinib for Patients With Advanced Unresectable (Stage IIIc) or Distant Metastatic (Stage IV) BRAF V600E/K Mutation Positive Cutaneous Melanoma
Brief Title: Access Study of Trametinib for Subjects With Advanced Unresectable (Stage IIIc) or Distant Metastatic (Stage IV) BRAF V600E/K Mutation Positive Cutaneous Melanoma
Status: No longer available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 202105
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Melanoma
Keywords: melanoma; dabrafenib; trametinib; BRAF V600E/K mutation
MeSH Terms: conditions — Melanoma | interventions — trametinib; dabrafenib

INTERVENTIONS:
Drug: Trametinib — Trametinib will be provided as tablets containing 0.5 milligram (mg) or 2.0 mg of trametinib parent (present as the DMSO solvate). The starting dose of trametinib will be administered orally 2.0 mg, once daily (QD)
Drug: Dabrafenib — Dabrafenib is commercially available as capsules containing 50 mg or 75 mg as free base (present as the mesylate salt). Dabrafenib will be administered orally 150 mg, twice daily (BID).

SUMMARY:
This is a single arm open label, multicenter, non randomized, access study of trametinib for subjects with histologically confirmed cutaneous melanoma with a BRAF V600E/K positive mutation that is either advanced unresectable (stage IIIc) or distant metastatic (stage IV). Trametinib may be given as monotherapy or in combination since first line metastatic melanoma as per inclusion criteria. Subjects who received prior BRAF inhibitor may be included if they have not progressed under such treatment or if they have presented limited progression as per eligibility criteria. It is estimated that between 250 and 400 subjects with histologically confirmed cutaneous melanoma with a BRAF V600E/K positive mutation that is either advanced unresectable (stage IIIc) or distant metastatic (stage IV) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Provides signed and dated informed consent, with age at the time of consent >=18 years.
* Has histologically confirmed cutaneous melanoma BRAF V600E/K positive mutation either unresectable (stage IIIc) or distant metastatic (stage IV).
* Is not eligible for enrolment in any other ongoing relevant hypothesis testing clinical study for metastatic melanoma or, if eligible, is so geographically distant from a participating site that attending frequent clinic visits is not feasible.
* Has not participated in the following GSK sponsored clinical studies (COMBI-v: MEK116513, COMBI-d: MEK115306, COMBI-AD: BRF115532) for melanoma indication prior to participating in this open label access study.
* Is able to swallow and retain oral medication.
* For subjects with active brain metastases: the subject does not require or is ineligible for immediate local treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 and in stable clinical condition. NOTE: subject in rapidly deteriorating clinical condition prior to start of therapy should not be considered for this open label access study. ECOG 3 subjects may be included provided the subject is clinically stable on the investigator's judgement.
* Does not require treatment with another anti-cancer therapy while on this open label access study (except dabrafenib if in combination with trametinib).
* Does not require treatment with prohibited concomitant medications.
* Does not have any medical conditions or physical examination or clinical laboratory findings which, in the opinion of the investigator and/or GSK Medical Monitor, would put the subject at high risk for an adverse outcome.
* Where applicable, female subjects of childbearing potential must agree to use one of the contraceptive methods listed in the study protocol. These subjects must have a negative serum pregnancy test within 7 days prior to the first dose of trametinib, preferably as close to the first dose as possible, agree to use adequate contraception from the time of the pregnancy test, throughout the treatment period and for a total of 4 months following the last dose of treatment.
* For subjects enrolled in France: a subject will be eligible for inclusion in this study only if he is, either affiliated to or beneficiary of a social security category.

Exclusion Criteria:

* Subjects who have received prior therapy with a MEK or BRAF inhibitor. NOTE: However subjects may be eligible in the following cases: Subjects whose tumor has not progressed based on radiographic and clinical assessments. Such subjects may receive therapy with: trametinib in combination with dabrafenib (in case of an adverse event related to a previous BRAF or MEK inhibitor other than trametinib or dabrafenib and without cross-reaction anticipated, or if clinically indicated according to investigator judgement). Prior treatment (except trametinib and dabrafenib) should have been stopped for a period of 5 half lives or 28 days (whichever is shorter) before starting treatment of this study; trametinib monotherapy if the subject has benefited from a treatment with a BRAF-inhibitor without progression but cannot receive it anymore due to tolerability reason. Subjects who have met the criteria for disease progression may receive trametinib in combination with dabrafenib if: the disease progression was confirmed after a period of at least 6 months of clinical benefit (Response or Stable Disease) on monotherapy and if the progression was characterized by a limited radiographic progression in the absence of clinical signs and symptoms of progression. no treatment-related grade 4 AEs or any SAEs occurred during the last 4 weeks of treatment.
* Concurrent treatment with other systemic anti-cancer therapies is not allowed (except dabrafenib in combination with trametinib). Subjects who are currently being treated with another systemic anti-cancer therapy (e.g. chemo, immune, biologic, or targeted therapy) must discontinue use prior to initiation of treatment in this open label access study for a period of 5 half lives or 28 days (whichever is shorter).
* Presence of malignancy other than melanoma within 1 year of enrolment into this program or any malignancy with confirmed activating RAS mutation. Subject with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Note: Prospective RAS testing is not required. However, if the results of previous RAS testing are known, they must be used in assessing eligibility.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib or dabrafenib, or excipients or to dimethyl sulfoxide (DMSO).
* Current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* Current evidence of cardiovascular risk including any of the following: Left Ventricular Ejection Fraction (LVEF) < lower limit of normal (LLN); A QT interval corrected for heart rate using the Bazett's formula >=480 millisecond (msec); Clinically significant uncontrolled arrhythmias; Acute coronary syndromes (including myocardial infarction and unstable angina); Congestive heart failure >=Class II as defined by New York Heart Association.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- France (44):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Chambray-lès-Tours
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Pringy
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Pierre
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Thionville
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valence
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif